CLINICAL TRIAL: NCT03389880
Title: Patellar Denervation in Total Knee Arthroplasty With Patellar Resurfacing to Relieve Postoperative Anterior Knee Pain: a Randomized Control Trial
Brief Title: Comparative Study Between Patellar Denervation and Non-patellar Denervation in Total Knee Arthroplasty With Patellar Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COA 147/2560
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Patellar Denervation; Non-patellar Denervation; Patellar Resurfacing
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patellar denervation (Active Comparator)
  Interventions: Procedure: Total knee arthroplasty; Procedure: Patellar denervation
- Non-patellar denervation (Experimental)
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — A surgical procedure in which parts of the knee joint are replaced with artificial parts (prostheses)
Procedure: Patellar denervation — circumpatellar electrocautery with monopolar coagulation diathermy
  Arms: Patellar denervation

SUMMARY:
The purpose of this study is to compare the post-operative anterior knee pain (AKP) between patellar denervation and non-patellar denervation in total knee arthroplasty with patellar resurfacing

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee who were scheduled for a primary total knee arthroplasty

Exclusion Criteria:

* Valgus deformity
* History of inflammatory arthroplathy
* Previous fracture or open surgery on the same knee
* History of patellar instability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Change of post-operative anterior knee pain | Change from baseline Visual Analog Scale for anterior knee pain at 3 months, 6 months, and 12 months after surgery
  Visual Analog Scale for anterior knee pain (minimum 0, maximum 10) Do higher values represent a worse outcome

SECONDARY OUTCOMES:
range of motion of knee | Change from baseline range of motion of knee at 3 months, 6 months, and 12 months after surgery
  degree of motion of the knee after surgery
Knee Society and Knee Society function score | Change from baseline Knee Society and Knee Society function score at 3 months, 6 months, and 12 months after surgery
  Knee Society and Knee Society function score (minimum 0, maximum 200)
New patellar score (Bartlett score) | Change from baseline new patellar score at 3 months, 6 months, and 12 months after surgery
  New patellar score or Bartlett score (minimum 0, maximum 30)
Oxford knee score | Change from baseline Oxford knee score 3 months, 6 months, and 12 months after surgery
  Oxford knee score (minimum 0, maximum 48)
patellar shift index | Change from baseline 3 months, 6 months, and 12 months after surgery
  The estimation of patellar position relative to the trochear
prevalence of anterior knee pain | Change from baseline prevalence of anterior knee pain at 3 months, 6 months, and 12 months after surgery
  Percent of anterior knee pain
activity of daily living | Change from baseline activity of daily living at 3 months, 6 months, and 12 months after surgery
  activity of daily living score (minimum 0, maximum 20)
post-operative complication | Number and type of post-operative complication at 3 months, 6 months, and 12 months after surgery
  Number and type of post-operative complication

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No